CLINICAL TRIAL: NCT03464994
Title: Prevalence of Ophthalmological Abnormalities in Children and Adults Suffering From Hereditary Ichthyosis
Brief Title: Ophthalmological Abnormalities in Hereditary Ichthyosis (ICHTYO-KERATO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Association for the development of research in Dermatology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/17/0067; 2017-A00605-48 (Other: ID-RCB)
Record Dates: First submitted 2017-11-18; First posted 2018-03-14 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ichthyosis
Keywords: Hereditary ichthyosis; keratoconus
MeSH Terms: conditions — Ichthyosis; Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ichthyosis patients (Other): patients presenting an Hereditary ichthyosis, whatever form or ongoing therapy will have an ophthalmological examination.
  Interventions: Diagnostic Test: ophthalmological examination
- control population (Other): patient without ichthyosis disease and consulting an ophthalmologist for refractive surgery screening or systematic eye examination will have an ophthalmological examination
  Interventions: Diagnostic Test: ophthalmological examination

INTERVENTIONS:
Diagnostic Test: ophthalmological examination — * Refraction
  * Best corrected visual acuity
  * Intraocular pressure
  * Slit lamp examination with vital dye (Oxford grading)
  * Tear break-up time (TBUT)
  * Schirmer I testing
  * Specular (TMS-4 Tomey) and elevation (pentacam Oculus and Orbscan Bausch & Lomb) corneal videotopographies
  * Pachymetry
  * Questionnaires: Ocular surface disease index, quality of vision (visual analogic scale), and quality of life (NEI-VFQ25)
  * questionnaire about ichthyosis severity
  * questionnaire about life quality specifically for patient presenting ichthyosis

SUMMARY:
Presence/absence of subclinical keratoconus with corneal topographic abnormalities (skewed radial axes for forme fruste keratoconus, and inferior steepening for keratoconus suspect) on axial specular topography (TMS-4 Tomey), and elevation topographies: Pentacam (Oculus) and Orbscan (Bausch & Lomb).

DETAILED DESCRIPTION:
Background: Hereditary ichthyosis are rare genetic diseases characterized by an abnormal epithelial keratinization due to mutations in gene involved in skin barrier. Patients present with scales on the whole body. Recent classification basically distinguishes syndromic from non-syndromic forms. Ichthyoses are severe diseases with significant impact on quality of life, due to troublesome symptoms (pruritus, pain), lack of effective therapy and complications such as ophthalmological anomalies. Among ophthalmological abnormalities, some are well known, such as eyelid abnormalities, including ectropion, and sicca syndrome. Conversely, corneal abnormalities such as keratoconus are not or very partially described in ichthyosis. The keratoconus is characterized by a corneal thickening and bulging with progressive loss of vision that may require a corneal transplantation. Its prevalence is 0.05% in its symptomatic presentation but may reach 10% when considering subclinical keratoconus diagnosed on basis of corneal topographies. These forme fruste keratoconus or keratoconus suspect may remain subclinical or instead progress to severe keratoconus. Corneal collagen crosslinking has been shown to strengthen the cornea in order to halt progressive keratoconus, justifying the need for early screening. Keratoconus is a complex condition of multifactorial etiology. With regards to the pathophysiology of the keratoconus, some hypotheses incriminate the corneal epithelial differentiation that is similar to the epidermal differentiation altered in ichthyosis. This link between both dermatological and ophthalmological abnormalities is supported by clinical experience. It's was observed that ichthyosis patients have frequently a subclinical keratoconus. In clinical practice, ophthalmological abnormalities are not commonly investigated in ichthyosis patients and there are no data on prevalence in the literature. Furthermore, there are no guidelines on screening or therapy of ophthalmological abnormities in ichthyosis.

The purpose of this project is to demonstrate that the prevalence of subclinical keratoconus (including forme fruste keratoconus and keratoconus suspect) is higher in ichthyosis compared to healthy controls.

Descriptive analysis of the studied population for primary outcome: The proportion of patients with subclinical keratoconus (including form fruste keratoconus and keratoconus suspect) will be described in each study-group and compared between study-groups using Mac Nemar Test.

ELIGIBILITY:
Inclusion Criteria:

For ichthyosis population:

* Hereditary ichthyosis, whatever form or ongoing therapy.
* Parental permission for minors

For controls:

* Patients who consult an ophthalmologist for refractive surgery screening or systematic eye examination
* Parental permission for minors

Exclusion Criteria:

For both populations:

* Patient who cannot stay seated
* Wearing contact lens within the last 7 days
* No social security
* Past medical history of corneal or eye surgery or eye condition (glaucoma, uveitis, keratoconus, retinal diseases)
* Impossibility to fill the questionnaires

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Presence/absence of subclinical keratoconus | 10 mn
  Presence/absence of subclinical keratoconus with corneal topographic abnormalities (skewed radial axes for forme fruste keratoconus, and inferior steepening for keratoconus suspect) on axial specular topography (TMS-4 Tomey), and elevation topographies: Pentacam (Oculus) and Orbscan (Bausch & Lomb).

SECONDARY OUTCOMES:
Presence/absence of symptomatic keratoconus with irregular topographic maps | 10 mn
  Evaluation by corneal videotopographies
Presence/absence of an abnormality of corneal transparency | 10 mn
  Evaluated by the measurement of the refraction,
Presence/absence of sicca syndrome | 10 mn
  Examination with the slit lamp of eyelids and eyelashes
Evaluation of quality of vision | 10 mn
  -Ocular Surface Disease Index (OSDI) : Self administered form to evaluate the impact of dry eye on visual function : 12 questions rated from 0 (never) to 4 (all the time)
Quality of life for adults | 10 mn
  -Quality of life by the National Eye Institute Visual Function Questionnaire (NEI-VFQ) : Self-administered questionnaire witch incorporates a wider range of data in relation to quality of life related to vision. Each question leads to an answer that is either dichotomous (yes / no), or graduated in 3, 4.5 and 6 points. The score of each item is transformed from 0 to 100, and the average of the scores by domain is established.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette MAZEREEUW, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided